CLINICAL TRIAL: NCT04650295
Title: Non-Pharmaceutical Intervention for Cirrhotic Cramps Reduction: The NICCles Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elliot B. Tapper, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00185598
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Cirrhosis; Muscle Cramp; Ascites
Keywords: Liver disease; Nutrition; quality of life; sleep; non-pharmaceutical intervention
MeSH Terms: conditions — Fibrosis; Muscle Cramp; Ascites; Liver Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Household Remedy (Experimental)
  Interventions: Other: Household Remedy
- Tap Water (Placebo Comparator)
  Interventions: Other: Tap water

INTERVENTIONS:
Other: Household Remedy — If the participant experiences a muscle cramp one tablespoon (one sip) of the household product will be taken. The treatment phase of the study will be for 28 days.
  Arms: Household Remedy
Other: Tap water — If the participant experiences a muscle cramp one tablespoon (one sip) of tap water will be taken. The treatment phase of the study will be for 28 days.
  Arms: Tap Water

SUMMARY:
This clinical trial is evaluating the feasibility of using a non-pharmaceutical treatment to improve the symptoms and severity of muscle cramps in patients with cirrhosis.

Eligible participants will be randomized to the treatment arm or control group. The treatment phase of the study will last 28 days. Information about participants will be collected including surveys and assessments throughout the study. Please note that only the participants randomized to experimental intervention group (Household Remedy) will be told what the treatment is during the study period. At the conclusion of the study (time of the final follow-up assessments), all participants will be debriefed on the use of concealment in this study as outlined in the protocol regarding the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cirrhosis (criteria per protocol will be used)
* History of painful muscle spasms, cramps, or charley horses that come on while resting (they had to have happened 4 times in the past month and bother the participant)

Exclusion Criteria:

* Non-English speaking
* Unable or unwilling to provide consent
* History of liver transplant
* History of multiple sclerosis
* History of cerebral palsy
* History of stroke with paralysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Reduction in cramp severity after 28-days as measured by the Visual Analog Scale for Cramps | 28 days
  This is a scale that is numbered from 0 (means no cramps) to 10 (worst cramps imaginable).

SECONDARY OUTCOMES:
Number of cramp-days per person | 28 days
Number of days with cramp severity less than 5 on the Visual Analog Scale for Cramps | 28 days
  This is a scale that is numbered from 0 (means no cramps) to 10 (worst cramps imaginable).
Number of cramps during study | 28 days
Change in sleep quality based on the Pittsburgh Sleep Quality Index (PSQI) | baseline, 28 days
  This study uses one question from the Pittsburgh Sleep Quality Index (PSQI) in which the participants reply how their sleep quality during the past month has been. Responses include: Very Good (0), Good (1), Fair (2), Bad (3), and Very Bad (4) the higher the score the worse the quality of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Tapper, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No